CLINICAL TRIAL: NCT04115033
Title: Randomized Double-Blind Placebo-Controlled Trial: fMRI Assessment of Cranial Electrical Stimulation for Fibromyalgia in Veterans
Brief Title: Randomized Controlled Trial of CES for Fibromyalgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3227-W; 1IK2RX003227-01 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: Pain; Fibromyalgia; Magnetic Resonance Imaging; Cranial Electrical Stimulation; Myofascial Pain Syndromes; Veterans
MeSH Terms: conditions — Fibromyalgia; Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Cranial electrical stimulation (CES) using a FDA-approved device that uses earclip electrodes to deliver current through the earlobe. The stimulator is meant to stimulate branches of the cranial nerves via the external ear.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- True CES (Experimental): Veterans with fibromyalgia who meet study criteria and are randomized to the experimental group will receive standard therapy in addition to cranial electrical stimulation (CES), which involves transfer of current from the alpha-stim device using earclip electrodes. The intention of this FDA-approved device is to relieve pain, though data on its effectiveness is still limited. The treatments can be self administered by the participants. The rs-fcMRI evaluation of neural changes and assessment of clinical pain, function, and quality of life will be performed at the beginning and end of the study.
  Interventions: Device: Alpha-stim
- Sham CES (Sham Comparator): Veterans with fibromyalgia who meet study criteria and are randomized to the sham comparator group will receive standard therapy in addition to a CES device that does not deliver active electrical stimulation. The intention of this FDA-approved device is to relieve pain, though data on its effectiveness is still limited. The rs-fcMRI evaluation of neural changes and assessment of clinical pain, function, and quality of life will be performed at the beginning and end of the study.
  Interventions: Device: Alpha-stim

INTERVENTIONS:
Device: Alpha-stim — The device for both groups is the Alpha-stim, a FDA-approved device similar to the Military Field Stimulator (MFS/Neuro-Stim System), a cranial electrical stimulation (CES) device.
  Other Names: Alpha-stim, CES

SUMMARY:
Given recent increasing opioid-related deaths and evidence showing against the use of opioids for non-malignant chronic pain, there is growing need for non-narcotic pain management. Fibromyalgia is a difficult to treat chronic pain condition that is often treated with opioids despite existing evidence. The prevalence of fibromyalgia is increased among Veterans returning from the gulf war and is already a significant burden in senior Veterans who may have suffered with chronic pain for decades already. Many treatment options for fibromyalgia carry intolerable side effects. CES (Cranial Electrical Stimulation) is a FDA-approved, non-pharmacologic therapy that is currently utilized within the military and VA system, but sufficient evidence regarding its outcomes and neural mechanisms have not been adequately investigated. An understanding of its neural underpinnings and analgesic effects could lead to 1) improvements in pain management and quality of life, 2) cost-savings and 3) development of new techniques to address pain.

DETAILED DESCRIPTION:
RESEARCH PLAN: In the setting of the opioid epidemic, it is crucial to develop non-pharmacologic treatments for pain and biomarkers to accurately assess pain treatment outcomes. In the present investigation, the investigators assess a novel non-pharmacologic approach to chronic pain treatment in patients suffering from fibromyalgia (a notoriously difficult to treat pain syndrome), utilizing neuroimaging as a biomarker. Resting state functional connectivity MRI (rs-fcMRI), a specific neuroimaging technique, has emerged as a reliable research tool to objectively assess, understand, and predict clinical pain in syndromes such as fibromyalgia. Preliminary results reveal a trend towards improved pain and function with a FDA-approved, non-pharmacologic therapy - auricular Cranial Electrical Stimulation (CES) - over standard therapy control, correlating to altered network connectivity on rs-fcMRI. CES-related improvements continued through 12 weeks following the completion of treatment and correlated to changes in cross-network connectivity, which differed between groups. OBJECTIVE: The proposed CDA-2, a randomized, sham-controlled trial of auricular CES, evaluates 1) the clinical utility of CES for fibromyalgia as compared to sham placebo control, 2) short- and long-term CES-related neural changes visualized on rs-fcMRI and 3) the ability of rs-fcMRI to predict CES treatment response. HYPOTHESIS: True CES results in non-placebo-related short- and long-term pain and functional improvements that can be correlated with altered connectivity and predicted by baseline rs-fcMRI. METHODS: Fifty total subjects (male and female Veterans, age 20-60 years old) will be randomized to either sham (n=25) or true (n=25) auricular CES. Neuroimaging data, self-reported pain, and function will be assessed at baseline and at 1 and 12 weeks post-treatment to evaluate neural correlates of CES-related treatment. Subjects who meet study criteria will receive baseline assessments including rs-fcMRI, Defense and Veterans Pain Rating Scale (DVPRS) measures, PROMIS measures, arm curl, 30-s chair stand, handgrip strength tests, and baseline analgesic consumption. Subjects will be block-randomized, stratified based on gender, to either true or sham CES (series of 4, weekly) treatments and assessed for rs-fcMRI and functional changes at 1 and 12 weeks post-treatment. This study addresses the critical need to identify and understand neural correlates of pain and non-opioid pain management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male and female Veterans age 20-60 with a diagnosis of fibromyalgia as diagnosed by a clinician, by chart review, and by the most recent American College of Rheumatology 2010 criteria for the diagnosis of fibromyalgia.
* Subjects must self-report consistent, daily pain (greater than 5 on the VAS) >90 days.
* Subjects must have intact skin free of infection at the site of electrode placement.
* Subjects must be willing to participate and understand the consent.
* Subjects must be right-handed in order to provide consistency in brain structure and function.

Exclusion Criteria:

* Subjects must not be currently pregnant, since effects of fMRI and electrical current on the developing fetus are not well-known.
* Subjects must not have an implanted electrical device such as a vagal stimulator, pacemaker, or spinal pain pump, which are not compatible with MRI.
* Subjects must not have a history of seizures or neurologic condition that may alter the structure of the brain.
* Subjects must not have a history of drug abuse or severe, uncontrolled psychiatric illness such as schizophrenia or major depressive disorder with suicidal ideation.
* Subjects must not have psoriasis vulgaris or other skin conditions that may increase the risk of infection at the implantation site.
* Subjects must not have severe anxiety, claustrophobia, or other conditions that may prevent their ability to lie at rest in an MRI scanner. This will be determined after discussion with the patient regarding their own perceived ability to lie at rest in an MRI scanner without the use of additional sedating medications.
* Subjects must not introduce new medications or treatments for fibromyalgia symptoms during the course of the study to prevent confounding results.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Pain Change | baseline, 1 week following treatment, and 12 weeks following treatment completion
  For subjects with fibromyalgia, clinical pain will be assessed in both groups using the Defense Veterans Pain Rating Scale (DVPRS), a validated measurement tool for pain, as well as analgesic consumption. Clinical pain will be measured at baseline, 1 week following treatment, and 12 weeks following treatment completion in both groups. The DVPRS is a combination of several different pain scales including the VAS, verbal rating scale, FACES scale, and numerical rating scale. Measurements will be graded on a scale of 0-10 with 0 being "no pain" and 10 being "severe" or "worst pain."

SECONDARY OUTCOMES:
rs-fcMRI Connectivity Change | baseline, 1 week, and 12 weeks following treatment completion
  Neuroimaging using resting state functional connectivity magnetic resonance imaging (rs-fcMRI) will be performed at baseline, 1 week, and 12 weeks following treatment completion in both groups to determine the short and long-term effects of PENFS on fibromyalgia-related altered network connectivity.
Sit-to-stand | baseline, 1 week, and 12 weeks following treatment
  Tests of function (sit-to-stand, bicep curl, handgrip strength) will be performed in both groups at baseline, 1 week, and 12 weeks following treatment. The sit-to-stand test tests how many full sit-to-stands a subject can perform within a 30 second interval.
PROMIS Change | baseline, 1 week, and 12 weeks following treatment
  NIH Patient-Reported Outcomes Measurement Information System (PROMIS) measures (sleep, mood, global health, etc.) will be assessed using a validated survey created from independently validated NIH PROMIS survey questions in both groups at baseline, 1 week, and 12 weeks following treatment.
Bicep-curl | baseline, 1 week, and 12 weeks following treatment
  Tests of function (sit-to-stand, bicep curl, handgrip strength) will be performed in both groups at baseline, 1 week, and 12 weeks following treatment. The bicep curl tests how many full bicep curls with gender specific weights (8 pounds for male, 5 pounds for female) a subject can perform within a 30 second interval. Both arms will be tested.
Handgrip strength | baseline, 1 week, and 12 weeks following treatment
  Tests of function (sit-to-stand, bicep curl, handgrip strength) will be performed in both groups at baseline, 1 week, and 12 weeks following treatment. The handgrip strength test uses a dynamometer to gauge the pressure that a subject can apply with their handgrip. Both hands will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Woodbury, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Case report: Percutaneous electrical neural field stimulation in two cases of sympathetically-mediated pain — https://f1000research.com/articles/6-920

DOCUMENTS (1):
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT04115033/ICF_000.pdf